CLINICAL TRIAL: NCT03344523
Title: A Randomized, Double-blind, Multi-center Clinical Trial Prospectively Evaluating Iron Protein Succinylate Oral Solution in Treating Patients With Chronic Heart Failure and Iron Deficiency
Brief Title: Evaluating Iron Protein Succinylate Oral Solution in Treating Chronic Heart Failure and Iron Deficiency
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-ZX02
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Chronic Heart Failure; Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — iron protein succinylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard treatment + Iron succinylate (Experimental): 1 bottle orally, twice daily, take orally before meals
  Interventions: Drug: Iron protein succinylate oral solution; Other: standard treatment
- standard treatment + placebo (Placebo Comparator): 1 bottle orally, twice daily, take orally before meals
  Interventions: Other: standard treatment

INTERVENTIONS:
Drug: Iron protein succinylate oral solution — Iron protein succinylate oral solution
  Arms: standard treatment + Iron succinylate
Other: standard treatment — standard treatment

SUMMARY:
This study aims to evaluate the effect of standard heart failure therapy plus oral solution with protein succinylate iron compared to placebo on the primary end point of 6 minute walk distance at 24th week in patients with chronic ejection fraction reduction heart failure and iron deficiency.

DETAILED DESCRIPTION:
This clinical trial was designed as a multicenter, prospective, randomized, double-blind controlled study. Patients were randomly divided into one of two treatment groups:

Control group: standard treatment + placebo（1 bottle orally, twice daily, take orally before meals, duration of treatment 16-24 weeks）.

Test group: standard treatment + Iron protein succinylate oral solution (1 bottle orally, twice daily, take orally before meals, duration of treatment 16-24 weeks）.

Sample size calculation is according to the change of 6 Minute walk distance from the baseline at 24 weeks, it is estimated the mean difference between two groups is 20 meter, standard deviation 80 meter, statistical power 80%, type I error 0.05, follow up loss 15%，estimated total sample size 600.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent form;
2. Between 18 to 80 years old, male or female;
3. Patients with chronic ejection fraction reduction heart failure, has been accepted the medication recommended by the Guidelines for treatment of heart failure in China (2014) for at least 4 weeks (that comply with the following requirements): if there is no contraindications or intolerance, patients should receive the renin angiotensin aldosterone system inhibitors, B blockers, and no dose adjustment within 4 weeks (not including diuretics). For patients who do not follow the guidelines for the use and titration of the renin angiotensin aldosterone system inhibitor and B blocker drugs, the cause should be recorded;
4. LVEF< 40% (determined by Simpson method) (valid for one week before randomization);
5. NYHA heart function II-III Grade;
6. NT-proBNP>400pg/ml, it should be .900pg/ml at atrial fibrillation;
7. Upper limit of hemoglobin: women less than 120g/L, men less than 130g/L. Lower limit of hemoglobin: more than 90g/L for both men and women. Accompanied by Iron deficiency (iron deficiency is defined as serum ferritin<100ug/L, or serum ferritin between 100~300ug/L with transferrin saturation (Tsat) <20%);
8. Capable of 6 Minute walk test.

Exclusion Criteria:

1. Patients with significant bleeding: gastrointestinal bleeding, menorrhagia, history of gastrointestinal bleeding and no evidence of gastrointestinal disease healing;
2. History of oral iron supplementation and intolerance;
3. History of acquired iron overload;
4. Exclude if receiving erythropoietin, intravenous iron, transfusion therapy and oral iron (including iron contained in compound vitamins or other compound medicine) ≧75mg/day within 6 weeks before enrollment;
5. Patients in urgent need of blood transfusion;
6. VtaminB12 and/or folate deficiency, unless correctable; and Non-iron deficiency anemia;
7. Severe renal insufficiency（eGFR < 20ml/min/1.73m2, MDRD formula）, renal anemia; or history of kidney dialysis, need of kidney dialysis at present or in 6 months;
8. Chronic liver disease, cirrhosis, active hepatitis, transaminases (increase of alanine aminotransferase and aspartate aminotransferase 3 times above the normal upper limit. Total bilirubin 3 times higher than the normal upper limit);
9. Intestinal diseases which affect iron absorption such as inflammatory bowel disease and chronic pancreatitis;
10. Active infection;
11. History of syncope within 3 months, diagnosed as cardiogenic shock over the past 1 months;
12. Active myocarditis, constrictive pericarditis and other pericardial diseases;
13. Acute decompensated heart failure with unstable hemodynamics;
14. Symptomatic bradycardia or second or third-degree cardiac conduction block with no pacemaker installed;
15. Severe chronic obstructive pulmonary disease, pulmonary heart disease, severe pulmonary vascular disease, pulmonary hypertension caused by autoimmune diseases and any type of severe pulmonary hypertension;
16. Valvular heart disease and congenital heart disease without operation; hypertrophic cardiomyopathy, restricted cardiomyopathy, and other secondary cardiomyopathy;
17. Patients with malignancy;
18. Patients combined with other organ diseases such as hematopoietic system, nervous system, endocrine system like thyroid, and combined with psychosis;
19. There is uncontrolled hypertension, systolic pressure is greater than 180mmHg and/or diastolic pressure is greater than 110mmHg;
20. Heart rate ≥ 130 times/minute before randomization, or malignant ventricular arrhythmia affecting hemodynamic;
21. Neuromuscular disease, disability or other non-cardiac causes influencing the performance of 6 Minute walk test;
22. Occurred within 3 months: acute coronary syndrome, stroke, transient cerebral ischemic attack; cardiac, carotid artery or other major vascular surgery; percutaneous coronary intervention (PCI) or carotid artery angioplasty or coronary bypass surgery and other cardiac surgery; or scheduled for percutaneous intervention and surgery surgical treatment within 6 months;
23. Has been implanted pacemaker/defibrillator (CRT-P/D) of cardiac resynchronization therapy within 6 months, or the intention to implant a similar device within 6 months after randomization;
24. Has been received major surgery within 6 months prior to randomization, or intend to receive major surgical treatment within 6 months;
25. History of heart transplantation or waiting for transplantation or using a left ventricular assist device (LVAD) or a heart transplant intention (waiting for transplantation) or intend to use VAD over the next 6 months;
26. Nursing or pregnant women, or women of childbearing age without contraception, or patients planned pregnancy in 6 months;
27. History of major organ transplant (such as lung, liver, bone marrow, kidney)
28. Patients have been involved or to be involved in other clinical trials within one month;
29. Patients cannot understand the informed consent form or cannot make decisions or of poor compliance;
30. Patients judged as unsuitable for the study and life expectancy less than 1 year by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The change of 6 Minute walk distances | 24 week
  The change of 6 Minute walk distances compared to baseline after patients receiving 24 week treatment.

SECONDARY OUTCOMES:
Variety of overall status score（PGA）after patients receiving 24 week treatment | 24 week
Kansas City Cardiomyopathy Questionnaire (KCCQ) rating change after patients receiving 24 week treatment | 24 week
Change of 6 Minute walk distance after patients receiving 16 week treatment | 16 week
Change of blood NT-proBNP after patients receiving 24 week treatment | 24 week
Cardiovascular death or heart failure re-hospitalization after patients receiving 24 week treatment | 24 week
Comprehensive cause mortality after patients receiving 52 week treatment | 24 week
EQ-5D Questionnaire score after patients receiving 24 week treatment | 24 week
Change of NYHA grading after patients receiving 24 weeks treatment | 24 week

OTHER OUTCOMES:
Index change in hemoglobin, serum iron, ferritin and transferrin saturation, and the like patients receiving 24 week treatment | 24 week
Index change in left ventricular ejection fraction, left atrial diameter, left ventricular diameter, pulmonary artery pressure and diastolic function after patients receiving 24 week treatment | 24 week
Rehospitalization with heart failure after patients receiving 24 week treatment | 24 week
Heart failure mortality after patients receiving 24 week treatment | 24 week
Cardiovascular readmission rates after patients receiving 24 week treatment | 24 week
Cardiovascular mortality after patients receiving 24 week treatment | 24 week
Comprehensive due readmission rates after patients receiving 24 week treatment | 24 week
Comprehensive cause mortality after patients receiving 24 week treatment | 24 week
C Reactive protein level after patients receiving 24 week treatment | 24 week

IPD SHARING:
Plan to Share IPD: No